CLINICAL TRIAL: NCT03544775
Title: Impact of Anesthesiology Interventions on Postoperative Outcomes in Adult Patients Undergoing Ambulatory Shoulder Surgery
Brief Title: Impact of Anesthesiology Interventions on Postoperative Outcomes in Adult Patients Undergoing Shoulder Surgery
Status: Completed | Type: Observational
Sponsor: Ottawa Hospital Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: GMH2
Record Dates: First submitted 2018-05-08; First posted 2018-06-04 (Actual); Results first posted 2024-11-27 (Actual); Last update posted 2024-11-27 (Actual); Status verified 2024-11

CONDITIONS: Postoperative Complications
MeSH Terms: conditions — Postoperative Complications | interventions — Immunoglobulin A

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Isolated General Anesthesia: Ontario residents, aged 18 years and older, who have undergone elective ambulatory shoulder surgery in Ontario and have not had a nerve block identified using physician billing codes.
  Interventions: Procedure: Isolated General Anesthesia
- Peripheral Nerve Block: Ontario residents, aged 18 years and older, who have undergone elective ambulatory shoulder surgery in Ontario and have a nerve block identified using physician billing codes.
  Interventions: Procedure: Peripheral Nerve Block

INTERVENTIONS:
Procedure: Isolated General Anesthesia — No nerve block identified through physician billing codes
  Other Names: iGA
  Groups: Isolated General Anesthesia
Procedure: Peripheral Nerve Block — Nerve block identified through physician billing codes
  Other Names: PNB+GA
  Groups: Peripheral Nerve Block

SUMMARY:
This retrospective, population-based cohort study will evaluate the comparative effectiveness of peripheral nerve blocks on patient outcomes after ambulatory shoulder surgery in adults patients undergoing surgery in Ontario.

DETAILED DESCRIPTION:
First, investigators will validate health administrative data codes to demonstrate the accuracy of Ontario-wide anesthesia type and regional anesthesia interventions using a reference standard (Ottawa Hospital Data Warehouse data). Then, these validated exposures, in combination with validated outcome measures, will be used to examine the impact of anesthesia interventions on patient and health system outcomes for ambulatory shoulder surgery.

ELIGIBILITY:
Inclusion Criteria:

* Ontario residents
* Aged 18 years and older
* Elective ambulatory shoulder surgery performed in Ontario between April 2009 and December 2016.

Exclusion Criteria:

* Emergency Surgery
* If a patient undergoes multiple elective shoulder surgeries within the time period, only the first surgery will be included for any participant in the study period.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: This will be a retrospective, population-based, cohort study based in Ontario, Canada. Our study population will include all Ontario residents, aged 18 years and older, who have undergone elective ambulatory shoulder surgery. The study period extends from April 2009 to March 2016.
Sampling Method: Non-Probability Sample
Enrollment: 59644 (Actual)
Dates: Start 2009-04-01 (Actual); Primary Completion 2016-03-31 (Actual); Study Completion 2018-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel McIsaac, MD, MPH, Principal Investigator — Department of Anesthesiology and Pain Medicine, University of Ottawa, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Isolated General Anesthesia | Peripheral Nerve Block
Started | 28571 | 31073
Completed | 28571 | 31073
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Isolated General Anesthesia | Peripheral Nerve Block | Total
Number analyzed (Participants) | 28571 | 31073 | 59644
Age, Continuous [Mean (Standard Deviation); unit: years] | 51 (13) | 52 (12) | 51 (12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9343 | 10534 | 19877
  Male | 19228 | 20539 | 39767
Surgery Type [Count of Participants; unit: Participants]
  Shoulder arthroplasty or joint repair | 11657 | 11342 | 22999
  Rotator cuff repair | 16571 | 19607 | 36178
  Other shoulder repair | 343 | 124 | 467
Surgery Type [Count of Participants; unit: Participants]
  Arthroscopic | 20314 | 23584 | 43898
  Open | 8257 | 7489 | 15746
Neighbourhood Income Quintile [Median (Inter-Quartile Range); unit: Neighbourhood income quintile] — Neighborhood socioeconomic status of the participants is presented as income quintile (income quintile is a measure of neighbourhood socioeconomic status that divides the population into five income groups (from lowest income to highest income)). The scale is from 1-5 (income group quintile 1 (lowest), 2, 3, 4, 5 (highest)). The groups are based on where 20% of the population falls within each category and therefore values vary by year.
  Neighbourhood income quintile | 3 [2 to 4] | 3 [2 to 4] | 3 [2 to 4]
Rural [Count of Participants; unit: Participants] | 5343 | 4039 | 9382
Healthcare resource use [Count of Participants; unit: Participants]
  Hospitalization in the last year | 1657 | 1523 | 3180
  Emergency department visit in the last year | 12543 | 12181 | 24724

OUTCOME MEASURES:

1. Primary Outcome: Postoperative Death, Admission, Readmission or Emergency Department Visits
Description: Composite outcome of: 1) unplanned admissions on the day of surgery , 2) post-discharge emergency department visits within 7 days of surgery, 3) readmission within 30 days of surgery, and 4) death from any cause
Time Frame: Date of surgery to 7 days (ED visits) and 30 days (readmissions) after surgery or death date, whichever came first
Population: Primary analysis
Measure: Count of Participants; unit: Participants
Arm/Group | Isolated General Anesthesia | Peripheral Nerve Block
Number analyzed (Participants) | 28571 | 31073
Participants
  Unplanned admission | 1,784 | 1,132
  Readmission within 30 days | 85 | 98
  ED visits within 7 days | 1,779 | 1,732
  Composite outcome | 3,424 | 2,808

2. Secondary Outcome: Health System Costs
Description: Costs in Canadian dollars will be calculated using standardized patient-level costing algorithms.
Time Frame: Date of surgery to 7 days and 30 days after surgery or death date, whichever came first
Measure: Mean (Inter-Quartile Range); unit: Canadian Dollars
Arm/Group | Isolated General Anesthesia | Peripheral Nerve Block
Number analyzed (Participants) | 28571 | 31073
Canadian Dollars
  Cost after surgery (7 days) | 4,391 [3910 to 4836] | 4681 [4337 to 5066]
  Cost after surgery (30 days) | 4528 [4014 to 5019] | 4840 [4451 to 5258]

3. Secondary Outcome: Neurology Consultations or Diagnostics
Description: Occurrence of neurology consult and/or nerve conduction study
Time Frame: Date of surgery to 90 days after surgery or death date, whichever came first
Measure: Mean (Standard Deviation); unit: Visits
Arm/Group | Isolated General Anesthesia | Peripheral Nerve Block
Number analyzed (Participants) | 28,571 | 31,073
Visits
  Neurology consultations in the 90 days after surgery | 74 (0.3) | 92 (0.3)
  Nerve conduction studies in the 90 days after surgery | 235 (0.8) | 274 (0.9)

ADVERSE EVENTS:
Time Frame: AEs were not collected
Description: AEs were not expected or collected.
Arm/Group | Isolated General Anesthesia | Peripheral Nerve Block
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
There is risk of misclassification bias. Confounding bias may influence receipt of specific interventions and outcomes. We were unable to measure patient-reported outcomes. Cost were captured at the health system level, but were not adequately granular to capture operating room supplies. We did not have specifics of each nerve block technique that may impact nerve block.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No